CLINICAL TRIAL: NCT05471531
Title: Immunogenicity and Safety of Quadrivalent Influenza Vaccine Combined Immunization With 23-valent Pneumococcal Polysaccharide Vaccine in the Elderly Aged 60 Years and Above
Brief Title: Study on Combined Vaccination With Quadrivalent Influenza Vaccine and 23-valent Pneumococcal Polysaccharide Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-INF4-MA4002-JStz
Record Dates: First submitted 2022-07-13; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Influenza and Pneumonia
MeSH Terms: conditions — Influenza, Human; Pneumonia | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined immunization group (Experimental): 160 subjects received one dose of quadrivalent influenza vaccine and one dose of 23-valent pneumococcal polysaccharide vaccine on day 0.
  Interventions: Biological: Combined vaccination with quadrivalent influenza vaccine and 23-valent pneumococcal polysaccharide vaccine
- Non combined immunization group (Experimental): There were two subgroups in non combined immunization group,and 160 subjects in each subgroup.The non combined immunization subgroup 1 received one dose of quadrivalent influenza vaccine on day 0 and one dose of 23-valent pneumococcal polysaccharide vaccine on day 28.The non combined immunization subgroup 2 received one dose of 23-valent pneumococcal polysaccharide vaccine on day 0 and one dose of quadrivalent influenza vaccine on day 28.
  Interventions: Biological: Separate vaccination with quadrivalent influenza vaccine and 23-valent pneumococcal polysaccharide vaccine
- Safety group (Experimental): 2520 subjects were enrolled and received one dose of quadrivalent influenza vaccine and one dose of 23-valent pneumococcal polysaccharide vaccine on day 0.
  Interventions: Biological: Combined vaccination with quadrivalent influenza vaccine and 23-valent pneumococcal polysaccharide vaccine

INTERVENTIONS:
Biological: Combined vaccination with quadrivalent influenza vaccine and 23-valent pneumococcal polysaccharide vaccine — Quadrivalent influenza vaccine and 23-valent pneumococcal polysaccharide vaccine were manufactured by Sinovac Biotech Co., Ltd.The routine of administration is intramuscular injection into deltoid region.And the immunization schedule is one dose of quadrivalent influenza vaccine and one dose of 23-valent pneumococcal polysaccharide vaccine on day 0.
  Arms: Combined immunization group; Safety group
Biological: Separate vaccination with quadrivalent influenza vaccine and 23-valent pneumococcal polysaccharide vaccine — Quadrivalent influenza vaccine and 23-valent pneumococcal polysaccharide vaccine were manufactured by Sinovac Biotech Co., Ltd.The routine of administration is intramuscular injection into deltoid region.And the immunization schedule is one dose of quadrivalent influenza vaccine on day 0 and one dose of 23-valent pneumococcal polysaccharide vaccine on day 28 in subgroup 1,and one dose of 23-valent pneumococcal polysaccharide vaccine on day 0 and one dose of quadrivalent influenza vaccine on day 28 in subgroup 2.
  Arms: Non combined immunization group

SUMMARY:
This study is an open-label,single center phase Ⅳ clinical trial of combined immunization with quadrivalent influenza vaccine and 23-valent pneumococcal polysaccharide vaccine.The purpose of this study is to evaluate the safety and immunogenicity of combined immunization with quadrivalent influenza vaccine and 23-valent pneumococcal polysaccharide vaccine in the elderly aged 60 years and above.

DETAILED DESCRIPTION:
This study is an open-label,single center,phase IV clinical trial in the elderly aged 60 Years and above.The experimental vaccines were manufactured by Sinovac Biotech Co., Ltd. A total of 3000 subjects will be enrolled,the safety and immunogenicity of combined immunization were evaluated in 480 subjects,and the Safety observation of combined immunization was evaluated in the extended safety group, which included 2520 subjects.

ELIGIBILITY:
Inclusion Criteria:

* The elderly aged 60 and above;
* The subjects and/or guardians can understand and voluntarily sign the informed consent form;
* Proven legal identity.

Exclusion Criteria:

* Received any circulating seasonal influenza vaccine prior to enrollment;
* Have received any pneumococcal vaccine within 5 years;
* History of severe allergic reactions to vaccines (such as acute anaphylaxis, angioneurotic edema, dyspnea, etc.);
* History of uncontrolled epilepsy and other serious neurological disorders (e.g.transverse myelitis, Guillain-Barre syndrome, demyelinating disease, etc.)
* Fever,acute onset of chronic disease,severe uncontrolled chronic disease or acute disease at the time of vaccination;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2021-11-13 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Immunogenicity index of Geometric mean titer(GMT) of influenza HI antibodies | 28 days after combined vaccination
  GMT of influenza HI antibodies for each influenza strain at 28 days after combined vaccination .

SECONDARY OUTCOMES:
Immunogenicity index of the seroconversion rates of influenza HI antibodies | 28 days after combined vaccination
  Seroconversion rate of influenza HI antibodies for each influenza strain at 28 days after combined vaccination.
Immunogenicity index of Geometric Mean Increase (GMI) of influenza HI antibodies | 28 days after combined vaccination
  GMI of influenza HI antibodies for each influenza strain at 28 days after combined vaccination.
Immunogenicity index of seropositivity rates of influenza HI antibodies | 28 days after combined vaccination
  Seropositivity rates of influenza HI antibodies for each influenza strain at 28 days after combined vaccination.
Immunogenicity index of Geometric Mean Concentration (GMC) for 23 serotypes specificity of pneumococcal IgG antibody | 28 days after combined vaccination
  GMC for 23 serotypes specificity of pneumococcal IgG antibody at 28 days after combined vaccination.
Immunogenicity index-seroconversion rates for 23 serotypes specificity of pneumococcal IgG antibody | 28 days after combined vaccination
  Seroconversion rates for 23 serotypes specificity of pneumococcal IgG antibody at 28 days after combined vaccination.
Immunogenicity index-GMI for 23 serotypes specificity of pneumococcal IgG antibody | 28 days after combined vaccination
  GMI for 23 serotypes specificity of pneumococcal IgG antibody at 28 days after combined vaccination.
Geometric mean titer(GMT) of influenza HI antibodies | 28 days after a single injection of quadrivalent influenza vaccine
  GMT of influenza HI antibodies for each influenza strain at 28 days after a single injection of quadrivalent influenza vaccine.
Seroconversion rates of influenza HI antibodies | 28 days after a single injection of quadrivalent influenza vaccine
  Seroconversion rates of influenza HI antibodies for each influenza strain at 28 days after a single injection of quadrivalent influenza vaccine.
Geometric Mean Increase (GMI) of influenza HI antibodies | 28 days after a single injection of quadrivalent influenza vaccine
  GMI of influenza HI antibodies for each influenza strain at 28 days after a single injection of quadrivalent influenza vaccine.
Seropositivity rates of influenza HI antibodies | 28 days after a single injection of quadrivalent influenza vaccine
  Seropositivity rates of influenza HI antibodies for each influenza strain at 28 days after a single injection of quadrivalent influenza vaccine.
Geometric Mean Concentration (GMC) for 23 serotypes specificity of pneumococcal IgG antibody | 28 days after a single injection of 23-valent pneumococcal polysaccharide vaccine
  GMC for 23 serotypes specificity of pneumococcal IgG antibody at 28 days after a single injection of 23-valent pneumococcal polysaccharide vaccine.
Seroconversion rates for 23 serotypes specificity of pneumococcal IgG antibody | 28 days after a single injection of 23-valent pneumococcal polysaccharide vaccine
  Seroconversion rates for 23 serotypes specificity of pneumococcal IgG antibody at 28 days after a single injection of 23-valent pneumococcal polysaccharide vaccine.
GMI for 23 serotypes specificity of pneumococcal IgG antibody | 28 days after a single injection of 23-valent pneumococcal polysaccharide vaccine
  GMI for 23 serotypes specificity of pneumococcal IgG antibody at 28 days after a single injection of 23-valent pneumococcal polysaccharide vaccine.
Safety index-incidence of adverse reactions | Within 7 days after combined immunization
  Incidence of adverse reactions at 0~7 after combined immunization with quadrivalent influenza vaccine and 23-valent pneumococcal polysaccharide vaccine.
Safety index-Incidence of adverse reactions | Within 28 days after combined immunization
  Incidence of adverse reactions at 0~28 after combined immunization with quadrivalent influenza vaccine and 23-valent pneumococcal polysaccharide vaccine.
Incidence of adverse reactions after a single injection of quadrivalent influenza vaccine | Within 7 days after a single injection of quadrivalent influenza vaccine
  Incidence of adverse reactions at 0~7 after a single injection of quadrivalent influenza vaccine.
The incidence of adverse reactions after a single injection of quadrivalent influenza vaccine | Within 28 days after a single injection of quadrivalent influenza vaccine
  Incidence of adverse reactions at 0~28 after a single injection of quadrivalent influenza vaccine.
Incidence of adverse reactions after a single injection of 23-valent pneumococcal polysaccharide vaccine | Within 7 days after a single injection of 23-valent pneumococcal polysaccharide vaccine
  Incidence of adverse reactions at 0~7 after a single injection of 23-valent pneumococcal polysaccharide vaccine.
The incidence of adverse reactions after a single injection of 23-valent pneumococcal polysaccharide vaccine | Within 28 days after a single injection of 23-valent pneumococcal polysaccharide vaccine
  Incidence of adverse reactions at 0~28 after a single injection of 23-valent pneumococcal polysaccharide vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongkui Zhu, Master, Principal Investigator — Taizhou Center for Disease Control and Prevention
Locations (4):
- China (4):
  - Jingjiang Center for Diseases Control and Prevention, Taizhou, Jiangsu
  - Taizhou City Hospital of Traditional Chinese and Western Medicine, Taizhou, Jiangsu
  - Gaogang District Center for Disease Control and Prevention, Taizhou, Jiangsu
  - Xinghua Center for Disease Control and Prevention, Taizhou, Jiangsu